CLINICAL TRIAL: NCT05220618
Title: Feasibility and Preliminary Effects an Online Training to Increase the Specificity and Savoring of Positive Autobiographical Memories: a Randomized Controlled Pilot Study
Brief Title: Efficacy of an Autobiographical Memory Specificity and Savoring Training for the Reduction of Depressive Symptomatology
Acronym: PESCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rosa M. Baños Rivera, Professor of Psychology, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1612004
Record Dates: First submitted 2022-01-04; First posted 2022-02-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Training Group; Control Group

STUDY DESIGN:
Intervention Model Description: This is a pilot study with a mixed between-subject design (experimental condition that will receive the training, and control condition that will only receive the assessment) and within-subject (pre/post-training assessment and 2-week follow-up). Continuous assessments will also be used to longitudinally evaluate participants during the 14 days of training and the 14 days of follow-up.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PESCAR Training Group (Experimental): This group will receive an online two-week intervention to train the specificity and savoring of autobiographical memories. During the two-week intervention and the following two weeks, participants will complete continuous assessments (i.e. once a day) rate the their mood (positive and negative affect) as well as the level of positivity, specificity and savoring of positive memories recalled during practice session. For this study, we included continuous assessments to monitor essential project variables throughout the intervention (2 weeks; from Day 0 to Day 15) and then as a follow-up (2 weeks after; from Day 16 to Day 30).
  Interventions: Behavioral: Autobiographical Memory Specificity and Savoring Training: PESCAR
- Control Group (No Intervention): This group will receive no intervention to train the specificity of autobiographical memories. During two weeks (from Day 0 to Day 15), participants will complete continuous assessments (i.e. once a day) to monitor their positive and negative affect.

INTERVENTIONS:
Behavioral: Autobiographical Memory Specificity and Savoring Training: PESCAR — An autobiographical memory specificity and savoring training has been developed by authors, based on previous training within the frame of Cognitive Bias Modification Interventions (CBM-I; Barry et al., 2019; Hitchcock et al., 2017) and savoring interventions (Bryant et al., 2005; Hanson et al., 2023). The training group will receive a self-guided intervention, which consists of an initial session (lasting 20 minutes approximately) and two-week training, conducted online. Participants will be provided with an online platform for following the intervention in a self-guided modality. The first session aims to give information about autobiographical memory functioning, to train in specificity recall through concrete processing steps and to explain the functioning of the self-guided modality. Then, during the next two weeks, participants will use the online platform once a day for practising the recall of autobiographical memories during 10-15 min approximately.
  Arms: PESCAR Training Group

SUMMARY:
The effect of autobiographical memory specificity and savoring training on memory specificity, positive affect regulation, well-being and depression symptomatology

DETAILED DESCRIPTION:
The general objective of this study is to analyze the efficacy of an online-delivered Autobiographical Memory Specificity and SavoringTraining to increase the specificity of positive autobiographical memories, positive affect regulation strategies, well-being and to reduce depression symptomatology. It will be tested in two conditions (training group vs. control group) with low-to-moderate depressive symptomatology. It is hypothesized that the training group (over control group) will increase the specificity and positive affect regulation of autobiographical memories, and this will lead to a reduction of depressive symptomatology and increase of well-being.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 (following Serrano et al., 2007 recommendations)
* Deficit in memory specificity: scores on Autobiographical Memory Test (AMT) < (or equal) 70%
* Diagnosis of mild to moderate depression: scores on Patient Health Questionnaire (PHQ9) between 5 to 14

Exclusion Criteria:

* being currently under psychological treatment
* present any medical illness or physical, psychological and/or cognitive incapacity that could impede the participation
* Not having the necessary technological means, i.e. access to a mobile phone with internet connection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Autobiographical memory specificity. The Autobiographical Memory Test (AMT, Williams & Broadbent, 1986) | Screening for eligibility criteria; Change in AMT from pre- intervention (Day 0) to post-intervention (Day 15)
  AMT is the preferred measure to evaluate the degree of specificity of autobiographical memory. During the AMT application, nine verbal cue words of different valence (three positive, three negative and three neutral) will be presented to the participants to perform a recall task of specific personal memories (Dritschel et al., 2014). The specificity of the memories is scored by evaluators following specified criteria (Williams et al., 2007), and then, an overall estimate of the level of specificity of autobiographical memories can be calculated. The assessment will be conducted online, following previous works with the written version of the AMT (Takano et al., 2017). The spanish adaptation (Ros et al., 2018) has shown adequate psychometric properties in young and older populations.

SECONDARY OUTCOMES:
Depressive symptomatology. The Patient Health Questionnaire 9 (PHQ-9; Kroenke, Spitzer & Williams, 2001, Spanish adaptation Diez-Quevedo et al., 2001) | Change in PHQ-9 from pre- intervention (Day 0) to post-intervention (Day 15); Change in PHQ-9 from post- intervention (Day 15) to follow-up (Day 30)
  PHQ-9 is a nine-item self-report measure of depressive symptoms. Participants answer the statements using a four-point Likert scale (0= Not at all to 3=Nearly every day) (Kroenke, Spitzer & Williams, 2001). The Spanish version has shown comparable diagnostic validity to the original English version, presenting levels of 88% of sensitivity and 88% of specificity (Diez-Quevedo et al., 2001).
Savoring. Ways of Savoring Checklist (WOSC, Bryant & Veroff, 2007; Jose, Lim, & Bryant, 2012) | Change in WOSC from pre- intervention (Day 0) to post-intervention (Day 15); Change in WOSC from post- intervention (Day 15) to follow-up (Day 30)
  An abbreviated 19-item os WOSC assess the use of thoughts and behaviours that facilitate savoring by amplifying positive feelings (11 items; for example, "I thought about sharing the memory of this later with other people") and the use of thoughts and behaviours that inhibit savoring by dampening positive emotions (eight items; for example, "I told myself why I didn't deserve this good thing"). Participants indicated to what extent statements described their thoughts and behaviours during positive experiences over the past week (1 = definitely doesn't apply, 7 = definitely applies). Previous studies have reported good psychometric properties with αs = .85-.86 (Smith and Hanni, 2019).
Characteristics of positive memories recalled. (Continuous assessments) | Daily mood and characteristics of positive memories during intervention (From Day 1 to day 15).
  Continuous assessment involves repeated sampling of subjects' behaviours and experiences in real time and in their natural environments, minimizing recall bias, maximizing ecological validity and allowing the study of micro-processes that influence behaviour. Previous studies have demonstrated the utility and validity of this assessment strategy in a variety of clinical and subclinical contexts (Colombo et al., 2020a, b).For this study, participants will record on their smartphones pre- and post- practice session measures. Pre-practice, participants will rate their mood (i.e. level of positive and negative affect). Post-practice, participants will rate their mood, and characteristics of the memory (i.e. level of specificity and positivity) and the recalling process (i.e. level of savoring and quality of the memory recall). This measure will be taken once a day, everyday during intervention (14 days: From Day 1 to day 15) and at follow-up (14 days; from Day 16 to Day 30)
Positive and negative affect. The Positive and Negative Affect Scale (PANAS; Watson et al., 1988; Sandín et al., 1999) | Screening for eligibility criteria; Change in PANAS from pre- intervention (Day 0) to post-intervention (Day 15); Change in PANAS from post- intervention (Day 15) to follow-up (Day 30)
  A self-report measure consisting of two sub-scales that assess the person's positive and negative affect. Each scale is composed of 10 items, giving a total of 20 items on a 5-point Likert scale (1=not at all/very mild; 5=extreme). The PANAS is established as a scale to measure changes in mood with excellent psychometric properties in the general population in its Spanish version (Sandín et al., 1999). In addition, its reliability and validity has recently been evaluated in the assessment of people with emotional disorders. It has shown good to excellent internal consistency in both subscales (Cronbach's alpha for positive affect = 0.91; Cronbach's alpha for negative affect = 0.87).
Well-being. Mental Health Continuum Scale (MHC: Keyes, 2004; Echevarría et al., 2010) | Screening for eligibility criteria; Change in MHC from pre- intervention (Day 0) to post-intervention (Day 15); Change in MHC from post- intervention (Day 15) to follow-up (Day 30)
  MHC-LF is a multidimensional measure, composed of 14 items measuring emotional (3 items), social (5 items) and psychological (6 items) well-being. It assesses the frequency with which they felt a certain way during the last month. Psychometric analyses of the Spanish validation (Echevarría et al., 2010) showed that it was a scale with good psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Baños, Full Professor, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Conunidad Valencia, Spain

REFERENCES:
- [Background] Takano K, Mori M, Nishiguchi Y, Moriya J, Raes F. Psychometric properties of the written version of the autobiographical memory test in a japanese community sample. Psychiatry Res. 2017 Feb;248:56-63. doi: 10.1016/j.psychres.2016.12.019. Epub 2016 Dec 16. PMID 28013087
- [Background] Ros L, Romero D, Ricarte JJ, Serrano JP, Nieto M, Latorre JM. Measurement of overgeneral autobiographical memory: Psychometric properties of the autobiographical memory test in young and older populations. PLoS One. 2018 Apr 19;13(4):e0196073. doi: 10.1371/journal.pone.0196073. eCollection 2018. PMID 29672583
- [Background] Barry TJ, Sze WY, Raes F. A meta-analysis and systematic review of Memory Specificity Training (MeST) in the treatment of emotional disorders. Behav Res Ther. 2019 May;116:36-51. doi: 10.1016/j.brat.2019.02.001. Epub 2019 Feb 2. PMID 30776658
- [Background] Hitchcock C, Werner-Seidler A, Blackwell SE, Dalgleish T. Autobiographical episodic memory-based training for the treatment of mood, anxiety and stress-related disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2017 Mar;52:92-107. doi: 10.1016/j.cpr.2016.12.003. Epub 2016 Dec 21. PMID 28086133
- [Background] Colombo, D., Suso-Ribera, C., Fernández-Álvarez, J., Cipresso, P., Garcia-Palacios, A., Riva, G., & Botella, C. (2020). Affect Recall Bias: Being Resilient by Distorting Reality. Cognitive Therapy and Research, 44(5), 906-918. https://doi.org/10.1007/s10608-020-10122-3